CLINICAL TRIAL: NCT01742052
Title: A Phase II, Multicentre, Randomised, Double-blind,Parallel Group, Placebo-controlled, Dose-finding Study to Evaluate the Safety and Efficacy of Three Different Oral Doses of MT-1303 Administered for a Period of 24 Weeks in Subjects With Relapsing-remitting Multiple Sclerosis
Brief Title: Dose-finding Study of MT-1303
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-1303-E04
Record Dates: First submitted 2012-12-02; First posted 2012-12-05 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: relapsing-remitting multiple sclerosis; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MT-1303-Low (Experimental): MT-1303-Low Dose
  Interventions: Drug: MT-1303-Low
- MT-1303-Middle (Experimental): MT-1303-Middle Dose
  Interventions: Drug: MT-1303-Middle
- MT-1303-High (Experimental): MT-1303-High Dose
  Interventions: Drug: MT-1303-High
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-1303-Low
  Arms: MT-1303-Low
Drug: MT-1303-Middle
  Arms: MT-1303-Middle
Drug: MT-1303-High
  Arms: MT-1303-High
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objectives of the study are:

* To evaluate the effects of three oral doses of MT-1303 compared to placebo given for a period of 24 weeks in subjects with relapsing-remitting multiple sclerosis (RRMS) on MRI parameters
* To evaluate the safety and tolerability of three oral doses of MT-1303 compared to placebo given for a period of 24 weeks in subjects with RRMS.

ELIGIBILITY:
Inclusion Criteria:

* RRMS as defined by the revised McDonald criteria
* Evidence of recent MS activity defined as either:

  * at least one documented relapse in the previous 12 months, OR
  * a positive gadolinium (Gd)-enhanced MRI scan within 3 months prior to screening, OR
  * at least two documented relapses in the previous 24 months with a positive Gd-enhanced MRI scan within the previous 12 months
* Expanded Disability Status Score (EDSS) score ≥0.0 and ≤5.5 points.

Exclusion Criteria:

* Primary progressive, secondary progressive or progressive relapsing MS at screening
* Disease duration >15 years combined with an EDSS score ≤2.0
* Relapse of MS during the Screening Period
* History or known presence of other neurological disorders likely to render the subject unsuitable for the study
* History of any of a list of pre-defined cardiovascular diseases
* History or known presence of any significant central nervous system, infectious, metabolic, oncological, ophthalmological or respiratory system disease or illness likely to render the subject unsuitable for the study
* Previous exposure to any sphingosine 1-phosphate receptor modulator
* Receipt of a live vaccine or systemic corticosteroid use within 28 days prior to randomisation
* Previous treatment with beta-interferons or glatiramer acetate within 14 days prior to randomisation
* Previous treatment with intravenous immunoglobulin, plasmapheresis, certain immunosuppressants, lymphocyte-depleting therapy, total body irradiation or bone marrow transplantation
* Need, or likely need for, treatment with Class I or III anti-arrhythmic drugs or with heart-rate-lowering beta-blockers or calcium-channel blockers, or with any other drugs which can reduce the heart rate
* Evidence of significant anaemia, thrombocytopenia, leucopoenia or lymphocytopenia, renal or hepatic impairment
* Clinically significant electrocardiogram (ECG) findings.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 415 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The total number of MRI Gd-enhanced T1-weighted lesions | Weeks 24

CONTACTS AND LOCATIONS:
Locations (18):
- Research Site, Brussels, Belgium
- Research Site, Sofia, Bulgaria
- Research Site, Edmonton, Canada
- Research Site, Zagreb, Croatia
- Research Site, Prague, Czechia
- Research Site, Vantaa, Finland
- Research Site, Berlin, Germany
- Research Site, Budapest, Hungary
- Research Site, Roma, Italy
- Research Site, Kaunas, Lithuania
- Research Site, Katowice, Poland
- Research Site, Moscow, Russia
- Research Site, Belgrade, Serbia
- Research Site, Madrid, Spain
- Research Site, Basel, Switzerland
- Research Site, Kozyatagi, Istanbul, Turkey (Türkiye)
- Research Site, Kiev, Ukraine
- Research Site, London, United Kingdom

REFERENCES:
- [Background] Kappos L, Arnold DL, Bar-Or A, Camm J, Derfuss T, Kieseier BC, Sprenger T, Greenough K, Ni P, Harada T. Safety and efficacy of amiselimod in relapsing multiple sclerosis (MOMENTUM): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2016 Oct;15(11):1148-59. doi: 10.1016/S1474-4422(16)30192-2. Epub 2016 Aug 16. PMID 27543447